CLINICAL TRIAL: NCT02055755
Title: Wound Research Database With Clinical Decision Support for Patients With Diabetic Foot Ulcers
Brief Title: WEMR With Clinical Decision Support for Diabetic Foot Ulcers
Status: Withdrawn | Type: Observational
Why Stopped: PI departure
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13309-1
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2016-09

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetes; Wounds; Wound Healing; Diabetic Foot Ulcer; DFU; Clinical Decision Support
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this project to begin using a wound research database with clinical decision support features at Winthrop University Hospital. A research database is an electronic computer system that is used to collect patient information. Clinical decision support is the ability for a computer system to provide medical assistance to the doctor through alerts and recommendations based on the information entered. The investigators believe that use of a wound clinical decision support tool, much like a drug, will improve healing in patients diagnosed with Diabetic Foot Ulcers and ultimately lower the risk of death and illness caused by these wounds. In order to develop a useful clinical decision support tool, investigators first need to develop a large research database to determine the data points important for wound healing. The investigators will be using the data collected in this study for future research and publication. Data will be reviewed to answer questions important to diabetic foot ulcer healing and for the purpose of developing the clinical decision support alert system.

After providing informed consent, participants will be asked a series of questions related to their past medical history, and relevant wound data will be collected. Study staff will photograph the wound at baseline, and once per week until the wound is completely healed, or for a duration of six months.

Participants will be expected to return to Winthrop University Hospital for wound follow-up on a regular basis, or as determined by the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Diabetes Type I, or Type II
* Must have a break in the skin on the plantar aspect of foot, > 0.5cm2
* Willing and able to provide written Informed Consent

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients at Winthrop University Hospital diagnosed with a Diabetic Foot Ulcer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire relevant to wound healing | up to 6 months
  * How do different types of bacterial infections affect DFU healing?
  * Does informing the patient and their families about wound characteristics improve DFU healing?
  * Which treatment modalities are the most optimal for managing patients with complicated DFUs (e.g. ischemic, infected)?
  * How does providing the patient with an individualized data summary and photos of their wound affect wound healing?

SECONDARY OUTCOMES:
Develop new parameters for clinical decision support based on data collected in this study. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harold Brem, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- See also: Related Info — http://complexwoundhealing.org